CLINICAL TRIAL: NCT04629612
Title: Regional Anesthesia in Non-intubated Breast Surgery, a Randomized Controlled Trial
Brief Title: Regional Anesthesia in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-05-001B
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasms; Pain; Analgesia; Regional Anesthesia
Keywords: Analgesia nociceptive index; Surgical pleth index
MeSH Terms: conditions — Breast Neoplasms; Pain; Agnosia | interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional anesthesia (Experimental): Regional block applied according to surgical area
  Interventions: Procedure: Regional anesthesia
- No Regional anesthesia (No Intervention): No regional anesthesia applied

INTERVENTIONS:
Procedure: Regional anesthesia — Regional anesthesia such as paravertebral block, pectoral block, superficial cervical plexus block, etc applies according to institution protocol
  Arms: Regional anesthesia

SUMMARY:
There is a trend that breast surgery can be done with peripheral nerve blockade and intravenous sedation, which reduces the side effects of general anesthesia such as nausea and vomiting, intubation discomfort and postoperative pain. The distribution of breast nerves is complex. Common nerve block methods are paravertebral blocks and pectoral nerve blocks. By monitoring the patient's heart rate variability change and measuring the patient's parasympathetic tone, the analgesic drug can be administered according to the patient's individual differences to avoid insufficient or excessive analgesic dose. The aim of this proposal is a prospective randomized controlled clinical trial is designed to evaluate changes in analgesia nociception index (ANI), surgical pleth index (SPI), postoperative opioid demand, and pain scores between patients who received regional anesthesia and those without in breast surgery patients under non-intubated surgery.

DETAILED DESCRIPTION:
Anesthesia has three elements: immobility, painlessness, and amnesia. To achieve these three factors depends on the balance between multiple factors, so multiple parameters need to be used for evaluation. In terms of subcortical function, pain indexes such as analgesia nociception index, surgical pleth index, etc. can be used to evaluate. By monitoring the parameters and comprehensive evaluation during the operation, the patient's condition can be fully understood. Opioids act on the central nervous system, making the nerve response slow and analgesic The effect is good, but there are many side effects, such as nausea and vomiting, drowsiness, respiratory depression, constipation, endocrine disorders, etc., and the central nervous system is suppressed by opioids, but the surrounding tissues are still damaged, releasing inflammatory mediators, causing immune dysfunction. Therefore, it is necessary to suppress inflammation and reduce the use of opioids, but also to effectively relieve pain. Nerve blockade is a powerful tool for this purpose. Local anesthetics are applied next to the nerves of the wound so that the pain signal cannot be transmitted to the central nervous system, reduce inflammatory mediators, reduce acute and chronic pain.

Breast surgery can be completed by peripheral nerve blockade and intravenous sedation, which can reduce the side effects of general anesthesia such as nausea and vomiting, intubation discomfort and postoperative pain. The distribution of breast nerves is complex, from the superficial cervical plexus, brachial nerve plexus, and thoracic vertebral nerves. At present, the commonly used nerve blocking methods include spinal nerve block, thoracic muscle block, brachial nerve block, and superficial nerve block. Blocking methods such as the cervical plexus, studies have shown that peripheral nerve blockade can reduce the amount of opioid analgesics during surgery.

This research plan is to design a randomized clinical trial to observe changes in the analgesic injury index (ANI), surgical pleth index (SPI), intraoperative and postoperative opiate demand, pain index, etc. inpatients with or without regional anesthesia under non-intubated breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Breast neoplasm require surgical resection of tumor
* Surgical type: non-intubated breast surgery under intravenous anesthesia

Exclusion Criteria:

* Contraindication for regional anesthesia: coagulopathy, infection
* Previous breast surgery
* Body mass index > 40
* Chronic opioid use
* Allergy to intravenous and regional anesthesia agents: Propofol, remifentanil, bupivacaine

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — On biological representation
Enrollment: 120 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid use | From start of post operative care unit to discharge from post operative care unit, up to two hours
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent
Post-operative opioid use | Second to 12th hour postoperatively
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent
Post-operative opioid use | 12th to 24th hour postoperatively
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent
Post-operative opioid use | 24th to 36th hour postoperatively
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent
Post-operative opioid use | 36th to 48th hour postoperatively
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent
Post-operative opioid use | 48th to 60th hour postoperatively
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent
Post-operative opioid use | 60th to 72nd hour postoperatively
  Total dose of post-operative morphine, tramadol, meperidine, etc calculated as morphine equivalent

SECONDARY OUTCOMES:
Intra-operative opioid use | From start of induction to completion of surgery, total of 1-2 hours
  Total dose of intra-operative remifentanil
Intra-operative analgesia nociception index | From start of induction to completion of surgery, total of 1-2 hours
  Intra-operative measurement of analgesia nociception index, on a scale on 0-100, higher on the scale indicate higher parasympathetic tone
Intra-operative surgical pleth index | From start of induction to completion of surgery, total of 1-2 hours
  Intra-operative measurement of surgical pleth index, on a scale on 0-100, lower on the scale indicate higher parasympathetic tone
Post-operative nurse rated pain scale | Second postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 6th postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 12th postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 24th postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 36th postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 48th postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 60th postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level
Post-operative nurse rated pain scale | 72nd postoperative hour
  Post-operative measurement of nurse rated scale, on a scale on 0-10, higher the score indicate higher pain level

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No